CLINICAL TRIAL: NCT05267574
Title: An Open-label, Multi-centre Study to Evaluate the Long-term Safety and Tolerability of REN001 in Subjects With Primary Mitochondrial Myopathy (PMM)
Brief Title: An Open Label, Long Term Safety Study of REN001 in Primary Mitochondrial Myopathy Patients (Stride Ahead)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Parent study failed to show therapeutic effect
Sponsor: Reneo Pharma Ltd (Industry)
Responsible Party: Sponsor
Organization: OnKure, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REN001-202
Record Dates: First submitted 2022-02-24; First posted 2022-03-04 (Actual); Results first posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-04

CONDITIONS: Primary Mitochondrial Myopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- REN001 (Experimental): 100 mg once daily
  Interventions: Drug: REN001

INTERVENTIONS:
Drug: REN001 — Once daily dosing

SUMMARY:
This study is designed to evaluate the long-term safety and tolerability of REN001 administered once daily to subjects with PMM due to mitochondrial DNA mutations (mtDNA-PMM) or nuclear DNA mutations (nDNA-PMM). Subjects with mtDNA mutations will have previously completed Study REN001-201 or participated in Study REN001-101. Subjects with nDNA mutations who enroll in this study will be REN001- naïve.

DETAILED DESCRIPTION:
This study is designed to evaluate the long-term safety and tolerability of REN001 administered once daily to subjects with PMM due to mitochondrial DNA mutations (mtDNA=PMM) or nuclear DNA mutations (nDNA-PMM). Subjects with mtDNA mutations will have previously completed Study REN001-201 (which is referred to as the STRIDE study) or participated in Study REN001-101. Subjects with nDNA mutations who enroll in this study will be REN001- naïve.

Eligible subjects will be treated with REN001 100mg orally, once daily for 24 months. Following the baseline visit there are planned visits at at defined time points. A final follow-up telephone call will be made by the study centre to the subject approximately 30 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* mtDNA-PMM subjects: Completed treatment in STRIDE or was participating in Study REN001-101 when the study stopped due to the COVID-19 pandemic, and in the opinion of the Investigator and Sponsor had been compliant with the study requirements OR nDNA-PMM subjects: Subjects aged 18 years or older with known nuclear (nDNA) pathogenic variants with a major muscle phenotype consisting of objective myopathy with poor exercise tolerance. Proof of pathogenicity must be provided. Must be able to walk at least 100m in the screening 12MWT and the limitations in walk test must be primarily due to the energy deficit and not due to ataxia or any other condition. For subjects under 25 years old only: confirmation of bone growth plate closure by wrist radiograph.
* Have PMM which continues to be primarily characterized by exercise intolerance or active muscle pain.
* Willing and able to swallow the REN001 gelatin capsules.
* Concomitant medications (including supplements) intended for the treatment of PMM or other co-morbidities likely to remain stable throughout participation in the study where clinically possible.
* Signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
* Females should be either of non-child-bearing potential or must agree to use highly effective methods of contraception from baseline through to approximately 30 days after the last dose of study drug. Males with partners who are women of childbearing potential (WOCBP) must also use contraception from baseline through to 14 weeks after the last dose of study drug.

Exclusion Criteria:

* Anticipated to need a peroxisome proliferator-activated receptor (PPAR) agonist other than REN001 during the study.
* Intent to donate blood, or blood components during the study or within one month after completion of the study.
* Current drug dependency. Use of opiates/cannabis for medical reasons is acceptable with prescription evidence or at the Investigator's discretion.
* Current alcohol dependency.
* Any medical, psychiatric or laboratory condition that may increase the risk associated with study participation or interfere with the interpretation of study results and, in the judgment of the Investigator and Medical Monitor, would make the subject inappropriate for entry into this study.
* Pregnant or nursing female

Subjects with mtDNA mutations can enroll at STRIDE Week 24 visit, STRIDE-FU visit, after exiting from STRIDE or after exiting REN001-101 (UK only). Subjects enrolling after exiting from either of the 2 feeder mtDNA studies and all subjects with nDNA mutations will be required to fulfill additional exclusion criteria during their additional screening visit. This is required for the mtDNA-PMM subjects due to the gap in study drug treatment and period of time without study assessments. The additional exclusion criteria are:

1. Clinically significant kidney disease or impairment calculated as eGFR Grade 2 or above <60ml/min/1.73m2 using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) creatinine equation at Screening.
2. Clinically significant liver disease or impairment of AST or ALT Grade 2 or above (>2.5 x ULN), or Total bilirubin > 1.6 x ULN or >ULN with other signs and symptoms of hepatotoxicity at Screening.
3. Subjects with uncontrolled diabetes and/or a Screening HbA1c of ≥11%.
4. Evidence of significant concomitant clinical disease that may need a change in management during the study or could interfere with the conduct or safety of this study. (Stable well-controlled chronic conditions such hypercholesterolemia, gastroesophageal reflux, or depression under control with medication (other than tricyclic antidepressants), are acceptable provided the symptoms and medications would not be predicted to compromise safety or interfere with the tests and interpretations of this study.)
5. Subjects with a history of cancer. A history of in situ basal cell carcinoma in the skin is allowed.
6. Clinically significant cardiac disease and/or clinically significant ECG abnormalities such as 2nd degree heart block, symptomatic tachyarrhythmia or unstable arrhythmia (right bundle branch block, left fascicular block and long PR interval are not excluded) that in the opinion of the Investigator should exclude the subject from completing exercise tests.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2024-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grainne Gorman, MD, Principal Investigator — Newcastle Hospital NHS Foundation Trust
Locations (29):
- Australia (3):
  - Royal North Shore Hospital, St Leonards, New South Wales
  - PARC Clinical Research, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
- University Hospital Leuven, Leuven, Belgium
- Canada (2):
  - M.A.G.I.C. Clinic (Metabolics and Genetics in Calgary), Calgary, Alberta
  - Vancouver General Hospital, Vancouver
- Copenhagen Neuromuscular Center, Copenhagen, Denmark
- France (6):
  - Hôpital Roger Salengro, Lille, Hauts-de-France
  - Centre de Référence des Maladies Neuromusculaires, Angers
  - Hôpital Neurologique, Bron
  - Nice Teaching Hospital, Nice
  - Hôpitaux Universitaires Pitié Salpêtrière, Paris
  - CHU de Strasbourg- Hopital de Hautepierre, Strasbourg
- Germany (2):
  - University Hospital Bonn Clinic and Polyclinic for Neurology, Bonn
  - Medical Center of the University of Munich Friedrich Baur Institute at the Neurological Clinic and Polyclinic, Munich
- Hungary (2):
  - Semmelweis University Insitute of Genomics and Rare Disorders, Budapest
  - University of Pécs Clinical Centre, Pécs
- Italy (5):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS Neurophysiopathology Unit, Rome, Lazio
  - A.O.U Policlinico di Messina U.O.C Neurologia e Malattie Neuromuscolari, Messina, Sicily
  - IRCCS Institute of Neurological Sciences of Bologna, Bologna
  - Istituto Nazionale Neurologico Carlo Besta, Milan
  - U.O. di Neurologia - Neurofisiopatologia, Pisa
- Radboud Universitair Medisch Centrum, Nijmegen, Netherlands
- Centre for Brain Research Neurogenetic Clinic, Grafton, Auckland, New Zealand
- Spain (2):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitari i Politècnic La Fe, Valencia
- United Kingdom (3):
  - Queen Square Centre for Neuromuscular Diseases, London, Greater London
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, Tyne and Wear
  - Salford Royal NHS Foundation Trust, Salford

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | REN001
Started | 155
Completed | 0
Not Completed | 155

BASELINE CHARACTERISTICS:
Arm/Group | REN001
Number analyzed (Participants) | 155
Age, Customized [Count of Participants; unit: Participants]
  18-25 years | 7
  26-45 years | 53
  46-64 years | 78
  >= 65 years | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 148
  Unknown or Not Reported | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4
  White | 144
  Not Reported | 5
  Other | 2
Region of Enrollment [Number; unit: participants]
  North America | 5
  Europe | 133
  Australia | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Mild, Moderate, Severe TEAEs, TEAEs Leading to Study Discontinuation, All TEAEs and All TESAEs
Description: Number of participants with AEs and severity
Time Frame: Baseline through study termination, an average of 12.1 months
Measure: Number; unit: participants
Arm/Group | REN001
Number analyzed (Participants) | 155
participants
  Mild TEAEs | 68
  Moderate TEAEs | 50
  Severe TEAEs | 5
  TEAEs leading to study drug discontinuation | 1
  Total TEAEs | 123
  Total TESAEs | 12

2. Secondary Outcome: Absolute Values, Changes From Baseline, and Incidence of Potentially Clinically Significant Changes in Laboratory Safety Tests, Electrocardiograms, Supine Vital Signs, and Eye Assessments
Description: Number of participants
Time Frame: Study Termination
Reporting Status: Not Posted

3. Secondary Outcome: Change in Distance Walked During a 12 Minute Walk Test
Description: Distance walked in meters
Time Frame: Baseline to Month 24
Reporting Status: Not Posted

4. Secondary Outcome: Change in Modified Fatigue Impact Scale (MFIS) Score
Description: The MFIS is a 21-item scale to describe the impact of fatigue on physical, cognitive, and psychosocial functioning. The questionnaire includes 9 physical, 10 cognitive, and 2 psychosocial items with each item scored between 0=Never and 4=Almost Always
Time Frame: Baseline to Month 24
Reporting Status: Not Posted

5. Secondary Outcome: Change in Patient Global Impression of Severity (PGIS) Score
Description: The PGIS is a 2-item questionnaire to describe the severity of fatigue and muscle symptoms. Each item is scored as Absent, Mild, Moderate, Severe, or Very Severe
Time Frame: Baseline to Month 24
Reporting Status: Not Posted

6. Secondary Outcome: Change in Brief Pain Inventory (BPI) Score
Description: The BPI is a 15-item questionnaire to describe severity of pain and its interference on functioning. The questionnaire includes 4 pain severity items each scored between 0=No Pain and 10= Pain, and 7 pain interference items each scored between 0=Does not Interfere and 10=Completely Interferes
Time Frame: Baseline to Month 24
Reporting Status: Not Posted

7. Secondary Outcome: Change in Patient Reported Outcomes Measurement Information System (PROMIS) Short Form - Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue 13a Scores
Description: The PROMIS Short Form - FACIT Fatigue 13a is a 13-item questionnaire to describe fatigue and its impact upon daily activities and function. Each item is scored between 1=Not At All and 5=Very Much
Time Frame: Baseline to Month 24
Reporting Status: Not Posted

8. Secondary Outcome: Change in 36-Item Short Form Health Survey (SF-36) Score
Description: The SF-36 is a 36-item questionnaire to describe health status and quality of life. The questionnaire includes 8 domains (physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions). Items are scored, summed into domains, and transformed into a scale of 0-100
Time Frame: Baseline to Month 24
Reporting Status: Not Posted

9. Secondary Outcome: Change Work Productivity and Activity Impairment Questionnaire: Specific Health Problem (WPAI:SHP) Score
Description: The WPAI:SHP is a 6-item questionnaire to describe impairment in work and activities due to a certain disease. Items are scored, summed, and transformed into a scale of 0-100%
Time Frame: Baseline to Month 24
Reporting Status: Not Posted

10. Secondary Outcome: Change in Patient Global Impression of Change (PGIC) Score
Description: The PGIC is a 2-item questionnaire to describe the change in fatigue and muscle symptoms since starting the study. Each item is scored as Very Much Worse, Moderately Worse, Minimally Worse, No Change, Minimally Improved, Moderately Improved, or Very Much Improved
Time Frame: Baseline to Month 24
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 48 months
Description: Regular Investigator assessment
Arm/Group | REN001
All-Cause Mortality (participants affected / at risk) | 0/155
Serious Adverse Events (participants affected / at risk) | 12/155
Other Adverse Events (participants affected / at risk) | 123/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | REN001 (N=155)
Cardiac Failure (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Ventricular Fibrillation (Cardiac disorders) | 1
Cerebrovascular Accident (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Radiculopathy (Nervous system disorders) | 1
COVID-19 (Infections and infestations) | 1
Campylobacter gastroenteritis (Infections and infestations) | 1
Compression fracture (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Cataract (Eye disorders) | 1
Intestinal Pseudo-obstruction (Gastrointestinal disorders) | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | REN001 (N=155)
COVID-19 (Infections and infestations) | 25
Upper respiratory tract (Infections and infestations) | 10
Influenza (Infections and infestations) | 9
Constipation (Gastrointestinal disorders) | 8
Fatigue (General disorders) | 12
Headache (Nervous system disorders) | 17
Myalgia (Musculoskeletal and connective tissue disorders) | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9
Dry skin (Skin and subcutaneous tissue disorders) | 8
Vitamin D deficiency (Metabolism and nutrition disorders) | 8
Refraction disorder (Eye disorders) | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An Investigator shall not publish any data (poster, abstract, paper, etc.) without having consulted with the Sponsor in advance.

DOCUMENTS (2):
  • Study Protocol (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT05267574/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-24): https://cdn.clinicaltrials.gov/large-docs/74/NCT05267574/SAP_001.pdf